CLINICAL TRIAL: NCT03692715
Title: A Multicenter Randomized Controlled Trial Assessing the Efficacy of Antimicrobial Prophylaxis for Extracorporeal Shock Wave Lithotripsy on Reducing Urinary Tract Infection
Brief Title: Antibiotic Prophylaxis Before Shock Wave Lithotripsy
Acronym: APPEAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Urology and Epidemiology Working Group (Other Government)
Collaborators: University of Helsinki (Other); Helsinki University Central Hospital (Other); Western University, Canada (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); King Abdulaziz University (Other); Hospital Sao Luiz (Other); St. Petersburg State Pavlov Medical University (Other); University Hospital, Basel, Switzerland (Other); Tallaght University Hospital (Other); Tabriz University of Medical Sciences (Other); Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Kari Tikkinen, Professor of Urology, Clinical Urology and Epidemiology Working Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLUE
Record Dates: First submitted 2018-08-21; First posted 2018-10-02 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Ureteral Stones; Ureteral Calculi; Nephrolithiasis
Keywords: ureteral stones; ureteral calculi; shockwave lithotripsy
MeSH Terms: conditions — Ureteral Calculi; Nephrolithiasis | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will undergo central randomization, which will be accessed by phone or internet. Un-blinding will occur only once statistical analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ciprofloxacin (Experimental): Single dose oral or intravenous ciprofloxacin prior to shockwave lithotripsy
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): identical oral placebo if oral cipro was used, or intravenous saline alone in a blinded fashion if IV cipro was used prior to shockwave lithotripsy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Oral or intravenous ciprofloxacin prior to shockwave lithotripsy.
  Other Names: Cipro
  Arms: ciprofloxacin
Drug: Placebo — identical oral placebo if oral cipro was used, or intravenous saline alone in a blinded fashion if IV cipro was used prior to shockwave lithotripsy.
  Arms: Placebo

SUMMARY:
This is a two arm, double blind RCT comparing the use of a single dose ciprofloxacin prior to SWL to saline alone. The multicenter trial will be conducted with a pragmatic emphasis including both high volume and low volume sites internationally.

DETAILED DESCRIPTION:
This is a two arm, double blind randomized controlled trial (RCT) comparing the use of a single dose ciprofloxacin prior to shock wave lithotripsy (SWL) to placebo. The multicenter trial will be conducted with a pragmatic emphasis including both high volume and low volume sites internationally.

Eligibility criteria include patients older than 18 years presenting for SWL who do not meet one of the pre-defined exclusion criteria (outlined below).

Eligible patients will provide written informed consent. Patients will undergo central randomization, which will be accessed by phone or internet. Un-blinding will occur only once statistical analysis is complete.

Patients will undergo SWL using standard procedures at the participating center. Participants will asked to provide a pre-procedure study questionnaire, a modified International Prostate Symptom Score (IPSS) questionnaire and a urine sample for analysis prior to SWL and follow-up. Follow-up questionnaires and a requisition for urine culture will be provided in a pre-stamped, self-addressed envelope along with instructions to return both culture and questionnaires to their participating center at 7-14 days post-SWL. If the follow-up questionnaire has not been received by post-operative day 10 patients will receive a reminder phone call. A second envelope will be sent containing a requisition for urine culture and follow-up questionnaire when necessary.

Alternatively, if a 2 week follow-up is conducted at the participating site then data-forms can be completed and collected at that time. In the event that a urine culture was not submitted 7 days post-operatively, one can be collected up to 14 days post-op. Additional clinical parameters such as presence of double J, stone characteristics and renal insufficiency will be recorded at the time of SWL by the dedicated research staff at the participating center. Data acquisition and occurrence of outcomes will be monitored continuously with scheduled audits.

Primary and secondary outcomes are outlined below.

The power calculation for this protocol was performed using Stata v.10.1 (StataCorp, College Station, TX). The investigators used the American Urological Association Best Practice Statement on antibiotic prophylaxis to estimate a 60% relative risk reduction with treatment arm. Therefore to achieve a power of 90% with a significance level of p<0.05, 661 patients will need to be recruited in each arm for a total of 1,322 patients. Accounting for 10% loss to follow-up, the total required will be 1454, or approximately 1500 patients. Assuming that 25% of patients screened will either refuse to be randomized or will meet one of the pre-defined exclusion criteria, a minimum of 2000 patients will need to be screened in order to randomize 1500 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 18 years presenting for SWL who do not meet one of the pre-defined exclusion criteria.

Exclusion Criteria:

* Pre-SWL urine analysis positive for nitrites
* Pre-SWL urine culture reveals >10e5 Colony Forming Unit/ml of bacteria (positive urine culture)
* Taking antibiotics for Urinary Tract Infection (UTI) or other cause
* Suspected struvite stone (based on previous stone analysis, or partial staghorn)
* Presence of nephrostomy tube
* Requiring cystoscopy and ureteral stent insertion on the day of SWL
* Presence of Foley catheter or patient on regular clean intermittent catheterization (CIC)
* Presence of urinary diversion (ie: ileal conduit)
* History of urosepsis prior to SWL
* Known allergic reaction to trial antibiotic
* Previous randomization in this trial
* In the opinion of the independent treating urologist, it is not in the patient's best interest to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1732 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Composite outcome including positive urine culture, symptoms of cystitis, pyelonephritis or urosepsis | 7-14 days post-shockwave lithotripsy
  The composite outcome with be assessed as a dichotomous variable. The presence of Positive post-SWL urine culture (≥ 10e5 Colony Forming Unit/ ml), with either one or more of symptoms of cystitis (defined as new onset burning sensation or pain with voiding, frequency, urgency), or pyelonephritis or urosepsis (hospital admission with fever ≥38.5 C) will be considered as an event.

SECONDARY OUTCOMES:
Bacteriuria defined as ≥ 100000 Colony Forming Unit/ml | 7-14 days post-shockwave lithotripsy
  Bacteriuria will be assessed as a dichotomous variable with presence of is ≥100000 Colony Forming Unit/ml will be considered as an event
Symptoms of cystitis defined as new onset burning sensation or pain with voiding, frequency, urgency | 7-14 days post-shockwave lithotripsy
  Symptoms of cystitis will be considered as a dichotomous variable with new onset burning sensation or pain with voiding, frequency, urgency will be considered an event
Pyelonephritis or urosepsis defined as Hospital admission with fever ≥38.5 Celsius | 7-14 days post-shockwave lithotripsy
  Pyelonephritis or urosepsis will be assessed as a dichotomous variable with Hospital admission with fever ≥38.5 Celsius will be considered as an event
Change in International Prostate Symptom Score (IPSS) total score (0-35, higher score indicates worse outcome) | 14 days post-shockwave lithotripsy
  Change in total value of IPSS score will be assessed as a continuous variable with a range from 0-35 with higher scores indicating more severe symptoms. This score is calculated by summation of individual component scores (0-5) across 7 domains
Individual components of International Prostate Symptom Score (0-7 per domain, with higher score indicating worse outcome) | 14 days post-shockwave lithotripsy
  Individual IPSS domains will be assessed as continuous variables and include incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Higher scores as considered as more severe symptoms
Pain scale determined on a range of 0-5 with higher score indicating worse outcome | 14 days post-shockwave lithotripsy
  Pain scale will be assessed as a continuous variable. The scale will be elicited by asking In the past week, how often have you had burning or discomfort with urination? Higher score is considered as more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kari AO Tikkinen, MD PhD, Principal Investigator — University of Helsinki; Philippe D Violette, MD CM, Principal Investigator — McMaster University
Locations (10):
- Hospital Sao Luiz, São Paulo, Brazil
- Canada (2):
  - Western University Hospital, London, Ontario
  - University of Sherbrooke, Sherbrooke, Quebec
- Helsinki University Hospital, Helsinki, Finland
- Universitas Indonesia - Cipto Mangunkusumo Hospital, Jakarta, Indonesia
- Tabriz University of Medical Science, Tabriz, Iran
- Tallaght University Hospital, Dublin, Ireland
- St Petersburg State Pavlov Medical University, Saint Petersburg, Russia
- King Abdulaziz University, Jeddah, Saudi Arabia
- Department of Urology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03692715/Prot_SAP_000.pdf
  • Informed Consent Form: Informed consent form Generic (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT03692715/ICF_001.pdf